CLINICAL TRIAL: NCT03691168
Title: Multi-center Observation of the Natural Course of Inherited Retinal Dystrophies
Acronym: RID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaodong Sun, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: Shanghai1stSXD
Record Dates: First submitted 2018-09-28; First posted 2018-10-01 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Inherited Retinal Dystrophies
Keywords: Inherited retinal dystrophies, Gene screen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Based on a clinical multi-center study of the natural course of inherited retinal dystrophies in Chinese population, screening fundus imaging indicators for patients with Chinese inherited retinal dystrophies, describing the clinical features of Chinese patients with inherited retinal dystrophies, and establishing a diagnosis of hereditary retinal diseases - Follow-up norms; establish a network-based multi-center diagnosis and follow-up platform; obtain a biological sample library of hereditary retinal diseases mainly in China. The research will further improve and enrich the genotype, phenotypic characteristics and natural course of Chinese inherited retinal dystrophies, in order to promote the clinical evaluation of clinical inherited retinal dystrophies and the standardization of genetic diagnosis. It is also the evidence for the best timing for future gene therapy, to obtain the best therapeutic effect, and to provide a theoretical basis for achieving precise treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with IRDs whose mutations have been identified
2. 4~70 years old
3. Complete 4 basic examinations of the eye: Corrective vision; fundus photography; OCT; ERG

Exclusion Criteria:

1. Has participated in other interventional treatment studies;
2. Patients with severe systemic diseases, mental dysplasia, mental illness;
3. Unable to accept eye examination patients;
4. Traumatic retinopathy, retinal inflammatory disease, paraneoplastic retinopathy, drug toxicity, and rare diseases such as diffuse unilateral subacute optic retinitis
5. At the initial visit, the patient's binocular vision is displayed as no light.
6. Both eyes have a history of internal eye surgery

Ages: 4 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with inherited retinal dystrophies
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 60 months
  A typical Snellen chart that if frequently used for visual acuity testing

CONTACTS AND LOCATIONS:
Overall Officials: XiaoDong Sun, PHD, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided